CLINICAL TRIAL: NCT05474794
Title: Diagnosis of Gastrointestinal Subepithelial Lesions Using a Novel Endoscopic Ultrasonography Imaging Technique
Brief Title: Detective Flow Imaging Endoscopic Ultrasonography in Subepithelial Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Principal Investigator, Carlos Robles-Medranda, Head of the Endoscopy Division, Instituto Ecuatoriano de Enfermedades Digestivas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IECED- 07202022
Record Dates: First submitted 2022-07-21; First posted 2022-07-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Leiomyoma; GIST
Keywords: Subepithelial lesion; detective flow imaging; Endoscopic Ultrasound-Guided Fine Needle Aspiration
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment A non-blinded, single center, non-randomized prospective, case control study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subepithelial lesions (Experimental): Patients with subepithelial lesions of the gastrointestinal (GI) tract (GISTs or leiomyomas) at EUS evaluation.
  Two interventions: EUS-DFI examination for the detection of slow flow vascularization in SELS. Then, CE-EUS for diagnosis confirmation.
  Interventions: Diagnostic Test: DFI-EUS; Diagnostic Test: CE-EUS

INTERVENTIONS:
Diagnostic Test: DFI-EUS — All patients enrolled having a confirmed histologic diagnosis of GIST or leiomyoma will undergo endoscopic ultrasound evaluation.
  First, the expert endoscopist will perform EUS-DFI examination for the detection of slow flow vascularization in SELS. Microvascularization EUS-Doppler evaluation will last between three and five minutes.
Diagnostic Test: CE-EUS — Immediately, after the first approach, CE-EUS (using Sulphur hexafluoride ultrasound contrast agent) will be performed for diagnosis confirmation. Sonovue will be administered intravenously in one (2.4 mL) or two administrations (4.8 ml), according to physician´s criteria, followed by an injected flush of 5 mL of sodium chloride solution (9 mg/mL).
  CE-EUS it will take around 5 minutes, with a total diagnostic approach around one hour.

SUMMARY:
Gastrointestinal stromal tumors (GIST) are the most common malignant subepithelial lesions (SELs) found in the gastrointestinal tract. The diagnosis and differentiation of these lesions from other subepithelial hypoechogenic tumors (i.e.as leiomyoma), is important as this may have an impact in the prognosis and treatment of either.

Due to GIST's notable features (vascularity and deep location), endoscopic ultrasound (EUS) is the first-line diagnostic approach. Based on this, three models (color-doppler EUS, power-doppler EUS, and e-FLOW EUS), are useful for real-time vascularity detection; however, these modalities are not helpful for fine and slow flow vessel detection. For overcoming this limitation, contrast-enhanced EUS (CE-EUS) is proposed as a first-line approach. Nevertheless, the use of contrast may be harmful, thus limited to some patients. To avoid contrast-related adverse events, a novel diagnostic method known as detective flow imaging endoscopic ultrasonography (DFI-EUS) has emerged. This technique detects fine vessels and slow flow without contrast. Despite the advantages of the latter, few studies have compared it with other diagnostic approaches in the evaluation and differentiation of SELs.

Hence, the investigators aim to evaluate the utility of DFI-EUS in the diagnosis of SELs (GIST and leiomyoma) by comparing it with CE-EUS.

DETAILED DESCRIPTION:
Subepithelial lesions (SELs) are a frequent finding on routine endoscopy (0.2%-3%), The importance of its diagnosis and management is based on its high risk of malignant transformation. According to literature, gastrointestinal stromal tumors (GIST) are the most common malignant SELs of the gastrointestinal tract. GIST appear as subepithelial lesions often covered by normal mucosa. For prognosis and treatment purposes, GIST should be differentiated from other benign submucosal hypoechogenic lesions such as leiomyoma, slow growing tumors, located preponderantly in the esophagus. The differential diagnosis between GISTs and leiomyoma is challenging because both can rise from the same second and forth muscular layers (muscularis mucosae and muscularis propria) and important because of the malignant potential of the former and consequently different management approach.

GISTs' diagnosis is approached by a combination of clinical signs and symptoms, laboratory tests and imaging techniques. Endoscopic techniques, such as esophagogastroduodenoscopy (EGD), is not useful to delineate the depth of invasion or subepithelial appearance of the lesions; also, conventional tissue acquisition through this modality is difficult when the tumor is not ulcerated. Due to this, EUS is considered critical for an accurate diagnosis, being the first-line diagnostic approach.

To date, color- doppler EUS, power doppler EUS, and e-FLOW EUS are EUS technologies that may be useful for observing vascularity in real time, but not for proper visualization of fine vessels and slow flow. On the other hand, contrast-enhanced EUS (CE-EUS) increases the detectability of vessels with high sensitivity yet holding the risk and limitations inherent to contrast administration.

To overcome diagnostic limitations, a new diagnostic method known as detective flow imaging endoscopic ultrasonography (DFI-EUS) has emerged. DFI-EUS detects fine vessels and low-velocity blood flow without the use of contrast agents. Despite its promising benefits, few studies have evaluated its advantages for the diagnosis and differentiation of GISTs. Only two studies have compared this technology against e-FLOW EUS, but in pancreatic tissue.

In the present study the investigators aim to evaluate the utility of DFI-EUS in the diagnosis of SELs (GIST and leiomyoma) by comparing it with CE-EUS.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our center with an indication of EUS for the evaluation of SELs
* Patients who authorized for DFI or CE-EUS.
* Written informed consent

Exclusion Criteria:

* Patients with contraindication for contrast agent administration.
* Any clinical condition which makes EUS-DFI or CE-EUS inviable
* Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of DFI-EUS in the identification of SELs | 1 day
  DFI effectiveness in the detection of vascularity in SELs will be assessed by the rates of identification of the intratumoral vessels. when compared with CE-EUS.
  Data from DFI and CE-EUS will be presented through a 2 x 2 contingency table.
Sensitivity and Specificity of DFI-EUS in the diagnosis of SELS | Up to 1 year
  Evaluate the sensitivity and specificity of DFI-EUS in the diagnosis of SELS. Data will be presented in percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas (IECED)
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas (IECED), Guayaquil, Guayas, Ecuador

REFERENCES:
- [Background] Yamashita Y, Yoshikawa T, Kawaji Y, Tamura T, Hatamaru K, Itonaga M, Ida Y, Maekita T, Iguchi M, Murata SI, Kitano M. Novel endoscopic ultrasonography imaging technique for visualizing microcirculation without contrast enhancement in subepithelial lesions: Prospective study. Dig Endosc. 2021 Sep;33(6):955-961. doi: 10.1111/den.13889. Epub 2020 Dec 23. PMID 33145842
- [Background] Yamashita Y, Yoshikawa T, Yamazaki H, Kawaji Y, Tamura T, Hatamaru K, Itonaga M, Ashida R, Ida Y, Maekita T, Iguchi M, Kitano M. A Novel Endoscopic Ultrasonography Imaging Technique for Depicting Microcirculation in Pancreatobiliary Lesions without the Need for Contrast-Enhancement: A Prospective Exploratory Study. Diagnostics (Basel). 2021 Oct 30;11(11):2018. doi: 10.3390/diagnostics11112018. PMID 34829364
- [Background] Casali PG, Blay JY, Abecassis N, Bajpai J, Bauer S, Biagini R, Bielack S, Bonvalot S, Boukovinas I, Bovee JVMG, Boye K, Brodowicz T, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dufresne A, Eriksson M, Fedenko A, Ferraresi V, Ferrari A, Frezza AM, Gasperoni S, Gelderblom H, Gouin F, Grignani G, Haas R, Hassan AB, Hindi N, Hohenberger P, Joensuu H, Jones RL, Jungels C, Jutte P, Kasper B, Kawai A, Kopeckova K, Krakorova DA, Le Cesne A, Le Grange F, Legius E, Leithner A, Lopez-Pousa A, Martin-Broto J, Merimsky O, Messiou C, Miah AB, Mir O, Montemurro M, Morosi C, Palmerini E, Pantaleo MA, Piana R, Piperno-Neumann S, Reichardt P, Rutkowski P, Safwat AA, Sangalli C, Sbaraglia M, Scheipl S, Schoffski P, Sleijfer S, Strauss D, Strauss SJ, Hall KS, Trama A, Unk M, van de Sande MAJ, van der Graaf WTA, van Houdt WJ, Frebourg T, Gronchi A, Stacchiotti S; ESMO Guidelines Committee, EURACAN and GENTURIS. Electronic address: clinicalguidelines@esmo.org. Gastrointestinal stromal tumours: ESMO-EURACAN-GENTURIS Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2022 Jan;33(1):20-33. doi: 10.1016/j.annonc.2021.09.005. Epub 2021 Sep 21. No abstract available. PMID 34560242